CLINICAL TRIAL: NCT03136666
Title: Single Dose Escalation Study to Investigate the Pharmacokinetics as Well as Safety and Tolerability of a Concomitant Administration of Nifedipne GITS and Candesartan Tablets Under Fasting Conditions in Healthy Male Subjects in an Open Label, Non-randomized, Sequential Design.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14026; 2010-018958-12 (EudraCT Number)
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — Nifedipine; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nifedipine + Candesartan cilexetil (Experimental): Coadministration of single doses of nifedipine and candesartan tablets
  Interventions: Drug: Nifedipine gastrointestinal therapeutic system (GITS) (Adalat LA, BAY a1040) + Candesartan cilexetil

INTERVENTIONS:
Drug: Nifedipine gastrointestinal therapeutic system (GITS) (Adalat LA, BAY a1040) + Candesartan cilexetil — Candesartan and nifedipine were administered together as loose combination with 240 mL non-sparkling water in the morning after a fasting period of at least 10 hours.

SUMMARY:
The objective of the study was to investigate the pharmacokinetics as well as safety and tolerability of a concomitant administration of nifedipine GITS and candesartan tablets under fasting conditions in healthy male subjects.

DETAILED DESCRIPTION:
* Treatment period 1: Single oral dose of 30 mg nifedipine GITS and 8 mg candesartan as loose combination (Treatment A)
* Treatment period 2: Single oral dose of 60 mg nifedipine GITS and 16 mg candesartan as loose combination (Treatment B)
* Treatment period 3: single oral dose of 60 mg nifedipine GITS and 32 mg candesartan as loose combination (Treatment C) Before any study drug administration in each treatment period, subjects were fasted from food for at least 10 hours. Subjects continued fasting until at least 4 hours after study drug administration. The wash-out phase between treatments was 5 days.

The blood collection period for pharmacokinetics after administration was 48 h. Afterwards, subjects were discharged from the ward. A safety follow-up visit was performed approximately 7 days after the last administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Age 30-55 years
* BMI 18.0-29.9 kg/m²
* Systolic blood pressure (SBP) ≥ 120 and ≤ 145 mmHg

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2010-06-07 (Actual); Study Completion 2010-06-07 (Actual)

PRIMARY OUTCOMES:
Overall summary of adverse events as a measure of safety and tolarability | 7 weeks
  Overview of treatment emergent adverse events and drug related adverse events, including information on severity as well as premature termination of study participation due to adverse events.
Safety related laboratory findings | 7 weeks
  Laboratory parameters were evaluated in terms of multiples of their upper limits of normal. Changes were considered relevant, if they were at least 1.5 times above the upper limit of normal.
Pharmacokinetic parameters: Maximum drug concentration in plasma after single dose administration divided by dose (mg) (Cmax/D) | 48 hours
Pharmacokinetic parameters: Area under the plasma concentration vs time curve from zero to infinity divided by dose (mg) (AUC/D) | 48 hours
Pharmacokinetic parameters: Maximum drug concentration in plasma after single dose administration (Cmax) | 48 hours
Pharmacokinetic parameters: Area under the plasma concentration vs time curve from zero to infinity after single (first) dose (AUC) | 48 hours

SECONDARY OUTCOMES:
Pharmacokinetic parameters: Maximum drug concentration in plasma after single dose administration divided by dose (mg) per kg body weight (Cmax,norm) | 48 hours
Pharmacokinetic parameters: Area under the curve divided by dose per kg body weight (AUCnorm) | 48 hours
Pharmacokinetic parameters: AUC from time 0 to the last data point (AUC(0-tn)) | 48 hours
Pharmacokinetic parameters: Time to reach maximum drug concentration in plasma after single (first) (tmax) | 48 hours
Pharmacokinetic parameters: Half-life associated with the terminal slope (t1/2) | 48 hours
Pharmacokinetic parameters: Mean residence time (MRT) | 48 hours
Pharmacokinetic parameters: Total body clearance of drug from plasma calculated after oral administration (apparent oral clearance) (CL/f) | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Wuppertal, North Rhine-Westphalia, Germany